CLINICAL TRIAL: NCT01277835
Title: Intravenous Lidocaine Infusion During VATS Procedures Reduces Postoperative Analgesic Requirements
Brief Title: Intravenous Lidocaine Infusion During Video-assisted Thoracic Procedures for Improved Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VATS-lidocaine
Record Dates: First submitted 2010-04-09; First posted 2011-01-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: video-assisted; thoracic surgery; VATS; lidocaine infusion; VATS procedures
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Infusion (Experimental)
  Interventions: Drug: Lidocaine Infusion
- Placebo (Placebo Comparator): Saline Infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Infusion — Infusion of lidocaine 3mg/min or 2mg/min during surgery
  Arms: Lidocaine Infusion
Drug: Placebo — Saline Infusion at same rate as experimental arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intravenous lidocaine infusion during a video-assisted chest surgery is effective in reducing the pain involved after the surgery. The hypothesis is that continuous lidocaine infusion during video-assisted thoracoscopic surgery (VATS) reduces morphine consumption and postoperative pain.

DETAILED DESCRIPTION:
Despite newer surgical techniques, many patients still experience moderate to severe postoperative pain after minimally invasive surgeries. Thoracoscopic surgeries are often associated with severe postoperative pain. To relieve the pain, potent narcotics have to be used, which have many side effects. Surgical patients would therefore benefit from an intra-operative analgesic regimen that is safe and effective, has minimal side effects and can reduce their postoperative narcotic requirements. Intravenous lidocaine has been shown previously to relieve cancer pain, chronic pain, and pain after other types of surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-75
* Scheduled for VATS procedure

Exclusion Criteria:

* Patients receiving antiarrhythmic therapy (Class Ia, Ib, Ic) within one week of surgery
* Patients on preoperative analgesic therapy within one week of surgery
* Patients with history of drug or alcohol abuse
* Patients who are allergic to lidocaine
* Contraindication to self administered morphine (unable to understand the PCA)
* Progression of the procedure to thoracotomy
* Patients who need postoperative mechanical ventilation
* Necessary major deviation from the intraoperative study protocol as per the discretion of the anesthesiologist in charge of the case
* Patients who are breastfeeding or pregnant
* Patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Verbal Rating Scale for pain with deep inspiration | Up to 48 hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about pain intensities with a deep inspiratory breath using the Verbal Rating Scale (0-10) at 8, 16, 24, 36, and 48 hours post-initiaition of patient-controlled analgesia.
PCA Morphine Consumption | Up to 48hrs post-initiation of patient-controlled analgesia
  Patient-controlled analgesia machines will be reviewed for the total morphine doses administered at 8, 16, 24, 36, 48 hours post-initiation of patient-controlled analgesia.
Number of PCA Morphine Requests | Up to 48hrs post-initiation of patient-controlled analgesia
  PCA machines will be reviewed for total number of PCA requests at 8, 16, 24, 36, 48 hours post-initiation of patient-controlled analgesia.
Verbal Rating Scale for pain at rest | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about pain intensities at rest using the Verbal Rating Scale (0-10) at 8, 16, 24, 36, 48 hours post-initiation of patient-controlled analgesia.

SECONDARY OUTCOMES:
Nausea | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about the side effect of nausea at 8, 16, 24, 36, 48 hrs post-initiation of patient-controlled analgesia.
Vomiting | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about the side effect of vomiting at 8, 16, 24, 36, 48 hrs post-initiation of patient-controlled analgesia.
Pruritus | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about the side effect of pruritus at 8, 16, 24, 36, 48 hrs post-initiation of patient-controlled analgesia.
Constipation | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about the side effect of constipation at 8, 16, 24, 36, 48 hrs post-initiation of patient-controlled analgesia.
Urinary Retention | Up to 48hrs post-initiation of patient-controlled analgesia
  Patients will be questioned about the side effect of urinary retention at 8, 16, 24, 36, 48 hrs post-initiation of patient-controlled analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ong, MD FRCPC, Principal Investigator — University of Saskatchewan, Department of Anesthesiology, Perioperative Medicine, and Pain Management; Brian Taylor, MD, Study Director — Department of Anesthesiology, Perioperative Medicine, and Pain Management; Ashraf Salem, MD, Study Director — Department of Anesthesiology, Perioperative Medicine, and Pain Management; Mark Slovack, MD, Study Director — Department of Anesthesiology, Perioperative Medicine, and Pain Management
Locations (1):
- St. Paul's Hospital, Saskatoon, Saskatchewan, Canada